CLINICAL TRIAL: NCT05074901
Title: Acceptance and Efficacy of a Smartphone-based App Using a Conversational Agent to Monitor Health Status and/or Deliver Behavioral Intervention to Reduce Psycho-social Stress
Brief Title: Virtual Agents-based Digital Interventions to Improve Health
Acronym: KANOPEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bordeaux (Other)
Responsible Party: Principal Investigator, Pierre Philip, Professor, University of Bordeaux
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHUBX2020GSP0102
Record Dates: First submitted 2021-09-20; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Mental Disorder; Mental Stress; Insomnia; Depression; Anxiety
Keywords: e-health; embodied conversational agent; ecological momentary assessment; ecological momentary intervention
MeSH Terms: conditions — Mental Disorders; Stress, Psychological; Sleep Initiation and Maintenance Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Open populational trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital behavioral intervention (Experimental): Digital behavioral interventions to improve mood and decrease fatigue, sleep complaints and substance usage.
  Interventions: Behavioral: digital behavioral intervention
- e-diaries (No Intervention): Ecological momentary assessment based on e-diaries on a weekly basis to evaluate sleep/wake schedules, physical activity, substance usage and nutrition.

INTERVENTIONS:
Behavioral: digital behavioral intervention — interaction with a conversational agent to implement physical and cognitive programs
  Arms: digital behavioral intervention

SUMMARY:
KANOPEE is a free smartphone application providing screening, follow-up tools and autonomous digital interventions to lower psycho-social stress and its repercussions on sleep and behaviors in the general population.

Additionally, KANOPEE permits an adaptation of the intervention to the subject (i.e., an adapted waiting period, frequency, and content), enabling to perform innovative trial conditions.

The objective of this long-term study is to evaluate the efficacy of KANOPEE on users among the French general population exposed to psycho-social stress.

DETAILED DESCRIPTION:
KANOPEE was designed by sleep specialists and psychiatrists to propose autonomous interventions to improve sleep, physical activity and substance abuse ; aiming at lowering psycho-social stress's repercussions. The app provides weekly interactions with a virtual companion.

At each interaction, users answer standardized questionnaires (e.g., Insomnia Severity Index, Cigarette Dependence Scale) enabling to characterize users' health status (i.e;, the severity of the complaints) and evolution over time, and therefore provide adapted interventions based on the literature (e.g., digital Cognitive Behavioral Therapies, diaries, sleep hygiene recommendations, motivational interviewing).

The app is freely available to the general population in France, enabling very large sample size, and the possibility to perform non-randomized trials depending on the selected interventions by the users and the subject's group.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18 years old and over (the app is available for younger users but their data will not be analyzed)
* having downloaded the app
* having a smartphone Android or Iphone
* being located in France
* having accepted the electronic informed consent

Exclusion Criteria:

* having clicked on the "emergency button" (in the app, there is a warning message : this app is not for emergency situations. If you need an urgent psychological support, click here")
* having downloaded the app but without answering any questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2020-04-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep complaints | weekly, from the downloading of the app until two weeks after the end of the intervention
  measured by the Insomnia Severity Index (ISI), total score ranging from 0 to 28, higher score indicating higher sleep complaint.
Fatigue complaints | weekly, from the downloading of the app until two weeks after the end of the intervention
  measured by the Fatigue Severity Scale (FSS), total score ranging from 1 to 7, higher score indicating higher perceived fatigue.
Depression and anxiety complaints | weekly, from the downloading of the app until two weeks after the end of the intervention
  measured by the Patient Health Questionnaire 4 items (PHQ-4), total score ranging from 0 to 12, higher scores indicating higher depression or anxiety complaints.

SECONDARY OUTCOMES:
Total Sleep Time | daily, from the downloading of the app until two weeks after the end of the intervention
  calculated based on the sleep diary data, corresponding to the actual time slept (Time in Bed - Sleep Onset Latency - Wakefulness After Sleep Onset - Terminal Wakefulness) (in hh:mm:ss)
Sleep Efficiency | daily, from the downloading of the app until two weeks after the end of the intervention
  calculated based on the sleep diary data, corresponding to the percent of time in bed spent asleep (Total Sleep Time/Time in Bed * 100) (percentage)
Time In Bed | daily, from the downloading of the app until two weeks after the end of the intervention
  calculated based on the sleep diary data, time starting from the moment of intention to fall asleep and concluding with the final arising (in hh:mm:ss).
Sleep Onset Latency | daily, from the downloading of the app until two weeks after the end of the intervention
  calculated based on the sleep diary data, corresponding to the time it takes to fall asleep, starting from the moment of intention to fall asleep (in hh:mm:ss)
Wakefulness After Sleep Onset | daily, from the downloading of the app until two weeks after the end of the intervention
  calculated based on the sleep diary data, corresponding to the total amount of time awake during the night (in hh:mm:ss)
Number of Awakenings | daily, from the downloading of the app until two weeks after the end of the intervention
  calculated based on the sleep diary data, corresponding to the total number of time awakenings during the night (number from 0 to 15)
number of episodes of craving | daily, from the downloading of the app until two weeks after the end of the intervention
  self-reporting number of moment during a day when the user felt the irresistible need to consume a substance (e.g., tobacco, alcohol)
amount of substance usage | daily, from the downloading of the app until two weeks after the end of the intervention
  self-reporting number of substance (e.g., cigarette, drinks) consumed during a day

OTHER OUTCOMES:
application's acceptance | facultative questionnaire that user can fill up after any interaction with the app (thus weekly)
  measured by the Acceptability of E-health Scale (AES), total score ranging from 0 to 30, higher score indicating a better acceptance of the app

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Philip, Pr, Principal Investigator — University of Bordeaux
Locations (1):
- University of Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sagaspe P, Sanchez-Ortuno MM, Dupuy L, Pecune F, Coelho J, Micoulaud-Franchi JA, Levavasseur Y, de Sevin E, Chanteclair A, Philip P, Salles N. Perceptions and Effectiveness of a Fully Automated Brief Behavioral Insomnia Therapy, Delivered by a Virtual Companion, in Older and Young Adults. Innov Aging. 2024 Sep 24;9(2):igae086. doi: 10.1093/geroni/igae086. eCollection 2025. PMID 40206328